CLINICAL TRIAL: NCT02541006
Title: A Randomized, Parallel-group, Phase IV Study to Compare the Bronchodilator Efficacy of Tiotropium (18 µg Once Daily [od]) Delivered Via a DISCAIR With Tiotropium (18 µg od) Delivered Via a HandiHaler®, in Patients With Moderate-to-severe COPD
Brief Title: Comparison of 24 Hour Bronchodilator Efficacy of Tiotropium 18 mcg Delivered Via DISCAIR Versus SPIRIVA 18 µg Delivered Via HANDIHALER® in Patients With Moderate to Severe COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neu-21.12
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2013-11

CONDITIONS: COPD
Keywords: FEV1; FVC; AUC 0-24; bronchodilator efficacy; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tiotropium 18 mcg dry powder for inhalation (Experimental): Tiotropium 18 mcg dry powder for inhalation, one inhalation, once daily with the DISCAIR
  Interventions: Drug: Tiotropium 18 mcg
- SPIRIVA 18 mcg HANDIHALER (Active Comparator): Tiotropium 18 mcg dry powder capsul for inhalation one capsule once daily with the HandiHaler
  Interventions: Drug: Tiotropium 18 mcg

INTERVENTIONS:
Drug: Tiotropium 18 mcg — tiotropium 18 mcg once a day

SUMMARY:
The objective of this study is to compare the bronchodilator efficacy a of tiotropium inhalation via DISCAIR (18 mcg once daily) and SPIRIVA HANDIHALER® (18 mcg once daily) in patients with moderate to severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years and older with moderate to severe COPD diagnosis
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* Patients with established clinical COPD and severity defined as a post-broncodilator FEV1/FVC ratio of ≤0.70 and FEV1 ≤80 % of predicted normal at screening
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods
* Have no excacerbation within last 4 weeks
* Hava capability of communicate with investigator
* Accept to adapt the procedures of study protocol
* Signed and dated informed consent

Exclusion Criteria:

* History of hypersensitivity to anticholinergics
* Diagnosis of asthma
* History of alergic rinit and athopy
* Current or history of lung cancer
* Known symptomatic prostatic hypertrophy requiring drug therapy
* Known narrow-angle glaucoma requiring drug therapy
* Have experienced exacerbation of COPD or lower respiratory inflammatory disease requiring use of antibiotics, oral or parenteral corticosteroids (CS) within 4 weeks prior to screening visit and/or during run-in period
* Patients vaccinated with poored virüs vaccinate within 2 weeks prior to screening visit and/or during run-in period
* Patients with a recent history of myocardial infarction, acute ischemic cardiac disease or severe cardiac arrhythmia requiring drug therapy
* Women who are pregnant or lactating or are planning on becoming pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Median maximum change (ml) from baseline in Forced Expiratory Volume in One Second (FEV1) and Forced Vital Capacity (FVC) | prior to the first dose of randomised study medication. Then, 15 minutes (min), 30 min,1 hour (h),2h,3h,4h,6h,8h,12 h and 24 h post dose
Percantage (%) change from baseline in FEV1 and FVC | prior to the first dose of randomised study medication. Then, 15 minutes (min), 30 min,1 hour (h),2h,3h,4h,6h,8h,12 h and 24 h post dose
Standardized Area Under the Curve (AUC) Between Baseline (Pre-dose) and 24 Hours -Post-dose | Baseline FEV1 taken at visit 2 prior to the first dose of randomised study medication. Then, 15 minutes (min), 30 min,1 hour (h),2h,3h,4h,6h,8h,12 h and 24 h post dose
- Forced Expiratory Volume in One Second (FEV1) Area Under the Curve From 0 - 24h (AUC 0-24) Response | Baseline FEV1 taken at visit 2 prior to the first dose of randomised study medication. Then, 15 minutes (min), 30 min,1 hour (h),2h,3h,4h,6h,8h,12 h and 24 h post dose

SECONDARY OUTCOMES:
Time to onset of bronchodilator effect and maximum effect | 15 minutes (min), 30 min,1 hour (h),2h,3h,4h,6h,8h,12 h and 24 h post dose
Adverse Events | predose and up to 24 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Neutec Ar-Ge San ve Tic A.S, Study Director — Neutec Ar-Ge San ve Tic A.S Clinical Trial

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yildiz P, Bayraktaroglu M, Gorgun D, Secik F. Bronchodilator efficacy of 18 mug once-daily tiotropium inhalation via Discair(R) versus HandiHaler(R) in adults with chronic obstructive pulmonary disease: randomized, active-controlled, parallel-group, open-label, Phase IV trial. Int J Chron Obstruct Pulmon Dis. 2016 Nov 22;11:2859-2867. doi: 10.2147/COPD.S119114. eCollection 2016. PMID 27920513